CLINICAL TRIAL: NCT00002212
Title: Phase II Evaluation of Targretin Capsules in Patients With AIDS-Related Kaposi's Sarcoma
Brief Title: A Study of Targretin Capsules in Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 287A; L1069-21
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Anticarcinogenic Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Bexarotene

INTERVENTIONS:
Drug: Bexarotene

SUMMARY:
The purpose of this study is to see if it is safe and effective to give Targretin capsules to patients with AIDS-related Kaposi's sarcoma (KS).

DETAILED DESCRIPTION:
This is a multicenter, open-label study to evaluate the safety and efficacy of Targretin capsules in patients with AIDS-related KS. NOTE: The daily dose may be reduced as necessary for toxicity management.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serum HIV antibody positive by ELISA.
* KS documented by biopsy (repeat biopsy is not required for entry if KS has been previously confirmed histologically and the histopathology report has been reviewed).
* A minimum of 6 mucocutaneous KS lesions, including at least 3 raised lesions, each of which has been present for at least 30 days or has a longest dimension of at least 10mm, and has not received prior local or topical therapy within 60 days of study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Concurrent, serious, uncontrolled infection including, but not limited to:
* Mycobacterium avium intracellulare or other mycobacterium infection; Pneumocystis carinii pneumonia; CMV retinitis or colitis; Toxoplasma brain abscess; Cryptococcal meningitis.
* Serious intercurrent illness or infection that would interfere with the ability of the patient to carry out the treatment program.
* Known allergy or sensitivity to retinoid class drugs.

Concurrent Medication:

Excluded:

* Local or topical therapy such as, but not limited to, Vitamin A, tretinoin (all-trans-retinoic acid), other retinoid class drugs, or intralesional (injection) therapy to any KS indicator lesion.
* Systemic anticancer chemotherapy, systemic anticancer hormonal therapy, and/or systemic anticancer immunotherapy.
* Systemic use of retinoid class drugs, beta-carotene compounds, or Vitamin A in doses greater than 15,000 IU (5,000 mcg) per day (equivalent to approximately 3 times the RDA) for any indication.
* Human chorionic gonadotropin.

Concurrent Treatment:

Excluded:

Radiotherapy, cryotherapy, photodynamic therapy, and/or laser therapy for any KS indicator lesion.

Prior Medication:

Excluded:

* Systemic treatment of KS within 30 days of study entry.
* Systemic treatment with either Vitamin A in doses greater than 15,000 IU (5,000 mcg) per day (equivalent to approximately 3 times the RDA) or other retinoid class drugs for any indication within 30 days of study entry.
* Previous local or topical therapy of any KS indicator lesion such as, but not limited to, Vitamin A, tretinoin (all-trans-retinoic acid), other retinoid class drugs, or intralesional (injection) therapy within 60 days of study entry.

Prior Treatment:

Excluded:

* Radiotherapy, cryotherapy, photodynamic therapy and/or laser therapy within 60 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Desert Univ School of Medicine, Palm Springs, California
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania